CLINICAL TRIAL: NCT07278999
Title: Effectiveness of Photobiomodulation, Er:YAG Laser, and Clobetasol in the Treatment of the Erosive Form of Oral Lichen Planus - a Randomized Clinical Trial.
Brief Title: Photobiomodulation, Er:YAG Laser, and Clobetasol in the Treatment of Oral Lichen Planus.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BNW/NWN/0052/KB1/124/25; BNW-1-151/N/5/K (Other Grant/Funding Number: Medical University of Silesia (Internal Grant))
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Oral Lichen Planus; Erosive Lichen Planus; Mucosal Lesions
Keywords: Oral lichen planus; lichen planus; laser; Er:YAG; Photobiomodulation therapy; steroids
MeSH Terms: conditions — Lichen Planus, Oral; Lichen Planus | interventions — Lasers, Semiconductor; Low-Level Light Therapy; Laser Therapy; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three independent treatment arms, each receiving a single intervention throughout the study period. The groups progress through the study simultaneously without crossover, allowing direct comparison of photobiomodulation, Er:YAG laser therapy, and topical clobetasol under a parallel design.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by an evaluator who is not involved in treatment delivery and will not have access to information identifying group assignment. Clinical measurements, lesion tracings, and photographic documentation will be coded before evaluation to maintain blinding. The assessor will review only de-identified data, ensuring that scoring of lesion size, mucosal features, and patient-reported measures is conducted independently of the intervention received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photobiomodulation (PBM) (Experimental): Participants in this arm receive photobiomodulation using a 635 nm diode laser delivered in continuous mode. Energy parameters follow a fixed protocol with 4 J/cm² fluence, 100 mW power, and 15 seconds per treatment point using a noncontact technique. Applications are performed twice weekly until complete epithelial healing or a maximum of eight sessions. This arm evaluates the regenerative and anti-inflammatory effects of PBM for erosive oral lichen planus.
  Interventions: Device: Photobiomodulation using 635 nm diode laser
- Er:YAG Laser Therapy (Experimental): Participants in this arm undergo Er:YAG laser treatment using pulsed energy with active cooling. The protocol applies controlled ablation of superficial mucosal lesions while minimizing thermal diffusion. Treatment is performed once weekly until full healing or a maximum of four sessions. This arm evaluates whether Er:YAG laser-assisted tissue removal supports faster healing and symptom reduction in erosive oral lichen planus.
  Interventions: Device: Er:YAG laser mucosal treatment
- Topical Clobetasol 0.05 percent (Experimental): Participants receive standard therapy with topical clobetasol propionate 0.05 percent. The medication is applied to clean, dry oral mucosa twice daily for thirty days following clinical guidelines for erosive oral lichen planus. This arm serves as the comparator for evaluating the effectiveness of laser-based treatments relative to established corticosteroid therapy.
  Interventions: Drug: Clobetasol propionate 0.05 percent topical application

INTERVENTIONS:
Device: Photobiomodulation using 635 nm diode laser — Photobiomodulation is delivered with a 635 nm diode laser in continuous mode at 100 mW, fluence 4 J/cm², and power density 0.2 W/cm². Each point is irradiated for 15 seconds using a noncontact technique with an 8 mm flat glass fiber tip and a 0.5 cm² spot size. Treatment points are spaced 2-3 mm apart over the lesion surface. Sessions are performed twice weekly until complete epithelial healing or for a maximum of eight sessions. This intervention aims to modulate inflammation and support mucosal repair in erosive oral lichen planus.
  Other Names: PBM laser therapy; Low level laser therapy (LLLT)
  Arms: Photobiomodulation (PBM)
Device: Er:YAG laser mucosal treatment — Er:YAG laser therapy is performed using pulsed energy at 50-80 mJ and 10 Hz (0.8 W) with a 300 µs pulse duration. Active cooling with water and air settings of 5/5 is applied. A flat fiber tip is used in a noncontact mode at a distance of approximately 3 mm from the lesion. The laser provides controlled superficial ablation of affected mucosal tissue to promote healing. Sessions occur once weekly until full epithelial recovery or for a maximum of four treatments. This intervention evaluates the therapeutic effect of Er:YAG laser-assisted tissue removal in erosive oral lichen planus.
  Other Names: 2940 nm laser therapy; Erbium:YAG laser
  Arms: Er:YAG Laser Therapy
Drug: Clobetasol propionate 0.05 percent topical application — Participants apply clobetasol propionate 0.05 percent directly to clean, dry oral mucosa twice daily for thirty days. The medication is used according to standard clinical practice for erosive oral lichen planus. The formulation serves as the active comparator to evaluate how laser-based treatments perform relative to conventional corticosteroid therapy. Participants are instructed to avoid eating, drinking, or rinsing for at least 30 minutes after application to ensure adequate mucosal contact.
  Other Names: Topical corticosteroid
  Arms: Topical Clobetasol 0.05 percent

SUMMARY:
This study aims to compare three treatment approaches for the erosive form of oral lichen planus, a chronic inflammatory condition that often causes pain, impaired oral function, and frequent relapses. Sixty adults with a confirmed diagnosis will be randomly assigned to photobiomodulation, Er:YAG laser therapy, or topical clobetasol, which serves as the current standard of care. The project investigates how effectively each method promotes healing of erosive lesions, reduces pain, improves oral functions such as chewing and swallowing, and prevents recurrence after treatment. Before enrollment, participants will undergo microbiological testing, tissue autofluorescence assessment, and histopathological confirmation. Treatment will follow strict protocols tailored to each therapy type, with PBM applied twice weekly, surgical laser once weekly, and clobetasol used twice daily for thirty days. Clinical outcomes will be measured using lesion size, standardized scoring systems, and patient-reported scales for pain and swelling. Follow up at one week, one month, and three months will document healing progress and relapse rates. Safety monitoring includes evaluation for infections and adverse reactions. The expected outcome is to determine which therapy provides the most effective, safe, and durable improvement. The study may offer evidence supporting laser based methods as alternatives that avoid the risks associated with long term steroid use.

DETAILED DESCRIPTION:
The study investigates three therapeutic approaches for managing the erosive form of oral lichen planus, a chronic inflammatory disorder of the oral mucosa characterized by persistent mucosal damage, pain, and the risk of recurrent symptoms. The erosive phenotype is clinically significant because it often leads to functional limitations, such as difficulty eating, impaired tolerance of removable prostheses, and reduced quality of life. Standard therapy relies primarily on potent topical corticosteroids, yet this approach is frequently limited by incomplete remission, recurrence after withdrawal, and the potential for local adverse effects, including mucosal atrophy and secondary candidiasis. For these reasons, alternative treatment modalities have gained increasing clinical interest, particularly those based on light-based therapies capable of modulating cellular processes or removing pathologic tissue with minimal collateral injury. Photobiomodulation and Er:YAG laser therapy represent two distinct applications of light energy. Photobiomodulation delivers low energy laser light that supports biological repair mechanisms, reduces inflammatory mediator activity, and enhances tissue regeneration without inducing thermal damage. Er:YAG laser treatment uses pulsed light at a wavelength strongly absorbed by water, which allows precise removal or gentle ablation of superficial diseased epithelium with limited thermal diffusion. This contributes to clean tissue surfaces and rapid re-epithelialization while preserving adjacent healthy mucosa. Although each method has been investigated in smaller clinical series, direct comparisons among photobiomodulation, Er:YAG laser therapy, and topical corticosteroids remain limited, especially when applied to the erosive variant of oral lichen planus. The study follows a parallel group design with allocation governed by block randomization to maintain balanced group sizes. Participants undergo diagnostic workup before allocation to ensure accurate confirmation of the disease subtype and to exclude other mucosal disorders with overlapping features. Autofluorescence imaging is used as part of the diagnostic process to support precise selection of biopsy site and to assist in distinguishing inflammation from dysplasia or other pathology. Only patients with disease confined to the oral mucosa and without evidence of systemic illness that could influence healing potential proceed to treatment. Interventions are performed using standardized protocols that reflect current best practices for each modality. Photobiomodulation is delivered with a diode laser operating under controlled parameters designed to stimulate repair pathways. The Er:YAG laser intervention uses short pulses with active cooling to ensure controlled ablation or superficial vaporization of the affected mucosa. The control arm uses a topical corticosteroid formulation routinely employed in dental medicine for erosive lesions, with instructions provided to support maximal mucosal contact time. During the treatment period, clinicians document changes in lesion characteristics using standardized measurement tools that allow objective quantification of mucosal surface area and morphological alterations. Photographic records supplement clinical scoring to ensure consistency across follow up visits. Pain severity and functional disturbances are captured with validated numeric scales, supporting a comprehensive evaluation that includes both clinical and patient centered components. Follow up assessments take place after treatment completion to examine the durability of mucosal healing. Given that erosive oral lichen planus often recurs, these visits are critical to understanding whether any modality provides sustained remission. Monitoring includes microbiological evaluation to detect any changes in colonization patterns, such as the emergence of yeast species that may influence treatment response or cause secondary symptoms. Safety oversight focuses on identifying adverse reactions such as erythema, mucosal irritation, delayed healing, dyschromia, or any unexpected tissue responses. Light based methods are generally regarded as safe when applied within established energy ranges, yet ongoing surveillance helps detect rare events or individual sensitivities. The protocol outlines criteria for early discontinuation when significant symptom exacerbation or other concerning findings emerge. This study is structured to deliver high quality comparative data that can guide clinical decision making when standard therapy is insufficient, poorly tolerated, or contraindicated. By evaluating three therapeutically relevant modalities, the study seeks to determine which approach most effectively promotes epithelial recovery, reduces symptom burden, and supports functional comfort. Its focus on recurrence patterns adds an important dimension, as durable improvement is often challenging to achieve in erosive oral lichen planus. The results may clarify the advantages of low level laser applications, the tissue conserving qualities of Er:YAG laser therapy, and the role of corticosteroids as a benchmark comparator. Photobiomodulation may demonstrate benefits related to noninvasiveness and absence of steroid related adverse effects. Er:YAG laser therapy may emerge as a precise alternative capable of controlling symptoms and accelerating healing while preserving nearby tissues. The study's methodology and extended observation window aim to support evidence based refinements to clinical protocols and promote therapeutic strategies aligned with patient comfort, safety, and long term disease control. The broader significance of the project lies in its potential to improve management of a chronic condition that has meaningful impact on daily activities and overall well being. By integrating structured clinical measurements, patient reported data, and advanced imaging methods, the study seeks to produce a comprehensive dataset that reflects contemporary standards in oral medicine research. The findings may pave the way for future work exploring predictors of treatment success, optimal energy settings for Er:YAG laser therapy, and potential combination approaches that incorporate both photobiomodulation and laser assisted tissue management.

ELIGIBILITY:
Inclusion Criteria:

* Be between 20 and 70 years old.
* Have histologically confirmed erosive or ulcerative oral lichen planus based on a biopsy.
* Have no active aerobic bacterial infection or oral fungal infection.
* Have had no treatment for OLP within the past 3 months.
* Provide written informed consent.

Exclusion Criteria:

* Systemic diseases or conditions such as uncontrolled diabetes (random glucose ≥200 mg/dl), cardiovascular failure, or a pacemaker.
* Autoimmune/connective tissue diseases such as lupus with positive ANA testing.
* Current or past cancer, graft-versus-host disease, or hematologic disorders (anemia, leukemia, lymphoma, bleeding disorders, hemophilia, von Willebrand disease).
* Enzymatic or metabolic disorders such as G6PD deficiency (favism) or porphyria.
* Viral hepatitis A, B, or C.
* Recent vaccinations (within the past 6 months).
* Use of medications known to trigger lichenoid reactions, including:
* Antihypertensives (beta-blockers, diuretics, ACE inhibitors, centrally acting agents).
* Oral antidiabetics (sulfonylureas).
* Metal-containing compounds (lithium, gold, arsenic, mercury).
* NSAIDs (e.g., ibuprofen).
* Antibiotics/chemotherapeutics (tetracyclines, sulfonamides).
* Pregnancy or breastfeeding (including up to 6 months post-lactation).
* Photosensitivity to UV light.
* Smoking more than 5 cigarettes per day.
* Lesions located adjacent to amalgam fillings or metal prosthetic restorations.
* Any degree of dysplasia on histopathology.
* Treatment for OLP within the last 3 months.
* Active oral fungal or bacterial infection at screening.
* Lack of consent to participate.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in erosive oral lichen planus lesion severity using the REA score | Baseline to 1 week after completion of assigned treatment
  Lesion severity will be measured using the REA scoring system, which evaluates the reticular (R), atrophic (A), and erosive (E) components of oral lichen planus. Each component is quantified from standardized lesion tracings and clinical measurements taken during oral examinations. Scores are calculated according to the protocol formula: REA = (R × 1) + (A × 1.5) + (E × 2). The change in total REA score from baseline reflects the therapeutic effect of each intervention on healing of erosive lesions.
Efficacy Index (EI) for overall treatment response | Baseline to 1 week after completion of assigned treatment
  The Efficacy Index (EI) quantifies overall clinical improvement using the formula defined in the study protocol:
  EI = [(total REA score before treatment - total REA score after treatment) ÷ total REA score before treatment] × 100 percent.
  EI will be used to categorize outcomes as complete healing, significant improvement, moderate improvement, mild improvement, or no improvement.
Improvement in pain intensity (NB) | Baseline to 1 week after completion of assigned treatment
  NB represents the percentage improvement in pain based on the Visual Analogue Scale (VAS). It is calculated using the formula:
  NB = [(VAS before treatment - VAS after treatment) ÷ VAS before treatment] × 100 percent.
  NB will classify improvement as complete, significant, moderate, mild, or absent.

SECONDARY OUTCOMES:
Change in lesion size measured in mm² | Baseline, 1 week, 1 month, and 3 months after treatment completion
  Lesion surface area will be measured using transparent millimeter-grid foil applied to the mucosal surface. Boundaries of each lesion will be traced and the total area calculated. Changes from baseline will be compared across treatment groups.
Change in pain intensity using the Visual Analogue Scale (VAS) | Baseline, 1 week, 1 month, and 3 months after treatment completion
  Pain will be assessed using a 0-10 VAS scale. Participants will report pain at baseline and at follow-up visits. Improvement will be quantified using the protocol-defined formula for pain reduction (NB).
Change in swelling or oral discomfort (subjective assessment) | Baseline, 1 week, 1 month, and 3 months after treatment completion
  Participants will evaluate swelling or discomfort on a 0-10 numeric scale. Improvement will be calculated using the protocol-defined formula (NO) to quantify reduction of symptoms after treatment.
Change in clinical grade using the Thonprasom scale (0-5) | Baseline, 1 week, 1 month, and 3 months after treatment completion
  Clinical severity of oral lichen planus will be evaluated using the Thonprasom grading system. Each lesion will be assigned a grade based on extent and morphology. Change in score over time will be used to assess therapeutic response.
Change in mycological status of oral mucosa | Baseline and 1 week after treatment completion
  Oral swabs will undergo mycological analysis to detect presence of Candida species before and after treatment. Results will identify whether any intervention increases or reduces fungal colonization or secondary infection risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves sensitive clinical information and the protocol does not include provisions for external data distribution. Data access is limited to the research team to protect participant privacy and confidentiality.

DOCUMENTS (1):
  • Study Protocol (2025-11-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT07278999/Prot_000.pdf